CLINICAL TRIAL: NCT02172222
Title: Relative Bioavailability of Multiple Doses BI 10773 50 mg and Linagliptin 5 mg After Concomitant Administration Compared to Multiple Doses of BI 10773 50 mg and Linagliptin 5mg Administered Alone to Healthy Male Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of BI 10773 and Linagliptin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.30
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Linagliptin

ARMS (2):
- Sequence ABC (Experimental): 1. Treatment A: BI 10773 once daily from day 1 to 5
  2. Treatment B: BI10773 and linagliptin once daily from day 1 to 7
  3. Treatment C: Linagliptin once daily from day 1 to 7
  Interventions: Drug: BI 10773; Drug: Linagliptin
- Sequence CAB (Experimental): 1. Treatment C: Linagliptin once daily from day 1 to 7
  2. Treatment A: BI 10773 once daily from day 1 to 5
  3. Treatment B: BI10773 and linagliptin once daily from day 1 to 7
  Interventions: Drug: BI 10773; Drug: Linagliptin

INTERVENTIONS:
Drug: BI 10773
Drug: Linagliptin

SUMMARY:
Study to investigate the relative bioavailability of BI 10773 and of linagliptin after concomitant multiple oral administration of 50 mg BI 10773 tablets and 5 mg linagliptin in comparison to 50 mg BI 10773 and 5 mg linagliptin given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers according to the following criteria:

  * Based upon a complete medical history and physical examination including vital signs (BP (blood pressure), PR (pulse rate)), 12-lead ECG (electrocardiogram) and clinical laboratory tests
* Age 18 to 50 years (inclusive)
* BMI 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation.

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 8
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 8

SECONDARY OUTCOMES:
tmax,ss (time from last dosing to the maximum measured concentration of each analyte in plasma at steady state) | up to day 8
Urine glucose excretion (UGE) | Pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 hours after the last dosing of each visit
Plasma DPP-4 (Dipeptidyl-peptidase 4) inhibition | 2 hours and 24 hours after last administration of study drug
Changes from baseline in physical examination | Baseline and within 5 days after last study drug administration
Changes from baseline in vital signs (blood pressure, pulse rate) | Baseline, day 1 and within 5 days after last study drug administration
Changes from baseline in 12-lead ECG (electrocardiogram) | Baseline and within 5 days after last study drug administration
Changes from baseline clinical laboratory tests | Baseline, day 1 and within 5 days after last study drug administration
Incidence of adverse events | Up to 56 days
Assessment of tolerability by investigator on a 4-point scale | Within 5 days after last study drug administration